CLINICAL TRIAL: NCT05066685
Title: Characteristics of Patients With Neovascular Age-related Macular Degeneration Enrolled in the Brolucizumab Patient Support Services Program
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRTH258AUS18
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Age-related Macular Degeneration (AMD)
Keywords: Primary plan,; AMD characteristics,; brolucizumab
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: All the particpants enrolled in the brolucizumab Patient Support Services (PSS) program
  Interventions: Other: All participants

INTERVENTIONS:
Other: All participants — All the particpants enrolled in the brolucizumab Patient Support Services (PSS) program

SUMMARY:
The study was a retrospective, cross-sectional, descriptive study of patients with wet AMD who enrolled in the brolucizumab Patient Support Services (PSS) program. Evidence was generated to describe their baseline demographic and clinical characteristics.

DETAILED DESCRIPTION:
The study was a retrospective, cross-sectional, descriptive study of patients with wet AMD who enrolled in the brolucizumab Patient Support Services (PSS) program.

PSS data was obtained from patients with wet AMD who enrolled in the program for the index period 10/10/2019 to 04/30/2020.

* Identification period of the index period: 10/10/2019 to 04/30/2020
* Index date: Date of enrollment in the PSS program
* Study Period: 10/10/2019 to 04/30/2020

ELIGIBILITY:
Inclusion Criteria:

* Patients were enrolled in the brolucizumab PSS program
* ≥19 years old

Exclusion Criteria:

• None

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included patients with wet AMD
Sampling Method: Probability Sample
Enrollment: 18457 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-09-25 (Actual)

PRIMARY OUTCOMES:
Number of patients with Primary plan type | Index date defined as the date of enrollment in the PSS program
  The primary plan type for patients with wet AMD enrolled in the brolucizumab patient support services program were reported. The primary Plan type include commercial, government or other insurance.

SECONDARY OUTCOMES:
Age | Index date defined as the date of enrollment in the PSS program
  Age information of patients enrolled in the brolucizumab PSS program was reported
Gender | Index date defined as the date of enrollment in the PSS program
  Gender information of patients enrolled in the brolucizumab PSS program was reported
Patient region (by state) | Index date defined as the date of enrollment in the PSS program
  Distribution of patients across US states
Provider region (by state) | Index date defined as the date of enrollment in the PSS program
  Number of providers and their distribution across US states
Insurance coverage | Index date defined as the date of enrollment in the PSS program
  The insurance coverage details for all the patients with wet AMD was reported
Number of patients with Secondary plan type | Index date defined as the date of enrollment in the PSS program
  The secondary plan type for patients with wet AMD enrolled in the brolucizumab patient support services program were reported. The secondary plan included commercial, government or other insurance
Disease Status | Index date defined as the date of enrollment in the PSS program
  The eye disease status of all the patients were reported. Disease status was categorized as Right eye, left eye, or bilateral

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, East Hanover, New Jersey, United States

REFERENCES:
- See also: Results for CRTH258AUS18 from the Novartis Clinical Trials Website — http://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17866